CLINICAL TRIAL: NCT04609423
Title: A Randomized, Parallel-group Treatment, Quadruple Masked, Two-arm Study, to Assess the Effectiveness of Cod Liver Oil Compared to Placebo in the Prevention of Covid-19 and Airway Infections in Healthy Adults
Brief Title: Cod Liver Oil for Covid-19 Prevention Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Arne Vasli Lund Søraas, Principal Investigator, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REK-172796
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Covid-19; Respiratory Tract Infections
Keywords: Cod liver oil; Vitamin D; n-3 LCPUFAs; SARS-CoV virus
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections | interventions — Cod Liver Oil; Vitamin D; RNA, Transfer; Corn Oil

STUDY DESIGN:
Intervention Model Description: A parallel-group treatment, two-arm study where participants are randomly assigned to cod liver oil or placebo (corn oil) in a 1:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, care providers, data collectors, outcomes assessors, and data analysts will be masked to the group assignment of each participant.
  Unmasking will be done after analysis of all primary endpoints and, preferably, also all secondary endpoints are completed.
  After unmasking the unmasked list will only be made available to study personnel needing this for conducting their tasks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cod liver oil (Experimental): supplementation for 6 months
  Interventions: Dietary Supplement: Cod liver oil
- Corn oil (placebo) (Placebo Comparator): supplementation for 6 months
  Interventions: Dietary Supplement: Corn oil (placebo)

INTERVENTIONS:
Dietary Supplement: Cod liver oil — 5 ml of cod liver oil as a source of 10 ug of vitamin D and 1.2 g of long-chained n-3 polyunsaturated fatty acids (DHA 0,6g and EPA 0,4g) per day for 6 months x 1 time/day together with the first meal of the day. 5ml of Cod liver oil also contains 250ug vitamin A and 10 mg vitamin E.
  Other Names: 10 ug of vitamin D and 1 g n-3 LCPUFA; Tran
  Arms: Cod liver oil
Dietary Supplement: Corn oil (placebo) — 5 ml of corn oil per day for 6 months x 1 time/day together with the first meal of the day
  Arms: Corn oil (placebo)

SUMMARY:
A randomized, parallel-group treatment, quadruple masked, two-arm study to assess the effectiveness of cod liver oil compared to placebo in the prevention of Covid-19 and airway infections in healthy adults.

In this study, the investigators will investigate whether daily cod liver oil can prevent Covid-19 infections and reduce the severity of such infections. The investigators will also examine whether cod liver oil prevents other airway infections in healthy adults.

DETAILED DESCRIPTION:
Preliminary evidence from literature and an ongoing study in the investigators' lab suggests that cod liver oil may prevent Covid-19 and complications of Covid-19. In the present study, the investigators will examine whether this is actually the case by randomizing volunteers to take cod liver oil or placebo (corn oil) during the winter months of 2020-2021. The investigators also aim to explore whether cod liver oil can prevent other respiratory tract infections, as well as explore and confirm already known health effects and possible new health effects, in particular rare adverse events associated with cod liver oil use.

Cod liver oil is a traditional source of vitamin A, D, and E and omega-3 fatty acids and the dose administered in the study will contain 250 ug vitamin A, 10 ug vitamin D, 10 mg vitamin E, and 1,2 g omega-3 fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Any person >18 years with a Norwegian Personal Identity Number

Exclusion Criteria:

* History of renal failure or dialysis, hypercalcemia, severe liver disease (cirrhosis), sarcoidosis or other granulomatous diseases (Wegener)
* Allergy to fish or corn oil.
* Pregnancy or planned pregnancy before summer 2021
* Vegan diet
* Age >75 years old at inclusion based on the Norwegian Personal Identity Number
* Difficulty in swallowing cod liver oil or other oils
* Previous Covid-19 disease
* For Caucasians only: Use of any supplement containing more than trace amounts of vitamin D or omega-3 fatty acids at inclusion (Vitamin D levels in non-Caucasians living in Norway are frequently low even among those self-reporting using dietary supplements). This criterion will be relaxed if too few participants volunteer for the study and only Caucasians that use cod liver oil or an equivalent dietary supplement (with omega 3 and vitamin D) more than 5-7 times per week will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47210 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with serious Covid-19 | 6 months
  The number of participants with first time SARS-CoV-2 positive nasopharyngeal and or pharyngeal swabs (or any other sample used for detection of current disease) analyzed by reverse transcriptase quantitative polymerase chain reaction (RT-qPCR) nucleic acid amplification test or antigen tests used by accredited Norwegian microbiology laboratories in the period from one week after the start of cod liver oil/placebo taking to the end of this period together with any of the following:
  A) Self-reported dyspnea and fever concurrent (within four weeks) with the positive test OR B) hospitalization caused by Covid-19 concurrent (within four weeks) with the positive test OR C) death where the Covid-19 infection was wholly or partly responsible as judged by the death certificate (see endpoint in the protocol)
Number of participants diagnosed with New Covid-19 | 6 months
  The number of participants diagnosed with first time SARS-CoV-2 positive nasopharyngeal and or pharyngeal swabs (or any other sample used for detection of current disease) analyzed by reverse transcriptase quantitative polymerase chain reaction (RT-qPCR) nucleic acid amplification test or antigen tests used by accredited Norwegian microbiology laboratories from one week after the start of cod liver oil/placebo taking.
Number of participants with negative SARS-CoV-2 test | 6 months
  Number of participants with an airway sample negative for SARS-CoV-2 (indicative of another airway infection).
  *Influenza virus (A and B), parainfluenzavirus (1,2,3), metapneumovirus, rhinovirus, coronavirus (non-SARS), Respiratory Syncytial virus, Haemophilus Influenzae, Moraxella Catharralis, Streptococcus Pneumonia, Beta-hemolytic streptococci, Mycoplasma pneumonia, Chlamydophila pneumonia, Enterovirus, Bordetella pertussis. The list can be expanded based on the analyses performed in Norwegian Microbiology laboratories.
Number of participants with self-reported airway infection | 6 months
  The number of episodes with any two of the following symptoms: fever, cough, nasal congestion or sore throat

SECONDARY OUTCOMES:
Number of participants hospitalized due to Covid-19 | 6 months
  Number of participants hospitalized wholly or partly caused by Covid-19.
Number of participants in Intensiv Care Unit (ICU) caused by Covid-19 | 6 months
  Number of participants with ICU care wholly or partly caused by Covid-19.
Number of participants with any admissions to hospital | 6 months
  Number of participants with any admissions to hospital based on the Norwegian Patient Registry data.
Infection with each of the mentioned pathogens | 6 months
  An airway sample positive for a respiratory pathogen* (either PCR or culture) in the period from one week after the start of cod liver oil/placebo taking to the end of this period.
  *Influenza virus (A and B), parainfluenzavirus (1,2,3), metapneumovirus, rhinovirus, coronavirus (non-SARS), Respiratory Syncytial virus, Haemophilus Influenzae, Moraxella Catharralis, Streptococcus Pneumonia, Beta-hemolytic streptococci, Mycoplasma pneumonia, Chlamydophila pneumonia, Enterovirus, Bordetella pertussis. The list can be expanded based on the analyses performed in Norwegian Microbiology laboratories.
Number of visits at GP for infections | 6 months
  Based on The Norwegian Reimbursement Database
Number of visits at GP | 6 months
  Based on The Norwegian Reimbursement Database

OTHER OUTCOMES:
Incidence of Cardiovascular disease | 6 months
  Based on self-reporting and Norwegian Registries
Incidence of Cardiovascular disease | 30 months
  Based on self-reporting and Norwegian Registries
Incidence of cardiovascular mortality | 6 months
  Based on self-reporting and Norwegian Registries
Incidence of cardiovascular mortality | 30 months
  Based on self-reporting and Norwegian Registries
Incidence of cancer | 6 months
  Based on self-reporting and Norwegian Registries
Incidence of cancer | 30 months
  Based on self-reporting and Norwegian Registries
Incidence of cancer mortality | 6 months
  Based on self-reporting and Norwegian Registries
Incidence of cancer mortality | 30 months
  Based on self-reporting and Norwegian Registries
All-cause mortality | 6 months
  Based on self-reporting and Norwegian Registries
All-cause mortality | 30 months
  Based on self-reporting and Norwegian Registries
Incidence of fracture of the hip or forearm | 6 months
  Based on self-reporting and Norwegian Registries
Incidence of fracture of the hip or forearm | 30 months
  Based on self-reporting and Norwegian Registries
Incident dementia | 6 months
  Based on self-reporting and Norwegian Registries
Incident dementia | 30 months
  Based on self-reporting and Norwegian Registries
Number of participants diagnosed with serious Covid-19 | 12 months
  The number of participants with first time SARS-CoV-2 positive nasopharyngeal and or pharyngeal swabs (or any other sample used for detection of current disease) analyzed by reverse transcriptase quantitative polymerase chain reaction (RT-qPCR) nucleic acid amplification test or antigen tests used by accredited Norwegian microbiology laboratories in the period from one week after the start of cod liver oil/placebo taking to the end of this period together with any of the following:
  A) Self-reported dyspnea and fever concurrent (within four weeks) with the positive test OR B) hospitalization caused by Covid-19 concurrent (within four weeks) with the positive test OR C) death where the Covid-19 infection was wholly or partly responsible as judged by the death certificate (see endpoint in the protocol)
Number of participants diagnosed with new Covid-19 | 12 months
  The number of participants diagnosed with first time SARS-CoV-2 positive nasopharyngeal and or pharyngeal swabs (or any other sample used for detection of current disease) analyzed by reverse transcriptase quantitative polymerase chain reaction (RT-qPCR) nucleic acid amplification test or antigen tests used by accredited Norwegian microbiology laboratories from one week after the start of cod liver oil/placebo taking.
Laboratory confirmed respiratory tract infection | 12 months
  An airway sample positive for a respiratory pathogen* (either PCR or culture).
  *Influenza virus (A and B), parainfluenzavirus (1,2,3), metapneumovirus, rhinovirus, coronavirus (non-SARS), Respiratory Syncytial virus, Haemophilus Influenzae, Moraxella Catharralis, Streptococcus Pneumonia, Beta-hemolytic streptococci, Mycoplasma pneumonia, Chlamydophila pneumonia, Enterovirus, Bordetella pertussis. The list can be expanded based on the analyses performed in Norwegian Microbiology laboratories.
Self-reported airway infection | 12 months
  The number of episodes with any two of the following symptoms: fever, cough, nasal congestion or sore throat
Number of participants with self-reported cod liver oil related adverse events | 12 months
  Number of participants with self-reported adverse events
Number of participants with cod liver oil related adverse events | 12 months
  Number of participants hospitalized for major diseases or death in the cod liver oil versus placebo group in Norwegian registries

CONTACTS AND LOCATIONS:
Overall Officials: Arne Søraas, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
IPD is complicated to share under the European General Data Protection Regulative, however, it is an aim of the study to make such data available within these regulations.

REFERENCES:
- [Derived] Brunvoll SH, Nygaard AB, Ellingjord-Dale M, Holland P, Istre MS, Kalleberg KT, Soraas CL, Holven KB, Ulven SM, Hjartaker A, Haider T, Lund-Johansen F, Dahl JA, Meyer HE, Soraas A. Prevention of covid-19 and other acute respiratory infections with cod liver oil supplementation, a low dose vitamin D supplement: quadruple blinded, randomised placebo controlled trial. BMJ. 2022 Sep 7;378:e071245. doi: 10.1136/bmj-2022-071245. PMID 36215222

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol version 1.2 without Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT04609423/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan version 1.0, signed (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT04609423/SAP_003.pdf